CLINICAL TRIAL: NCT04354857
Title: Qualitative and Quantitative Evaluation of Anosmia Over Time in Clinically Symptomatic Patients Tested for COVID-19 Infection
Acronym: Anosmie-COVID
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: IRB: 20.04.09
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: COVID-19
Keywords: anosmia; SARS-Cov-2
MeSH Terms: conditions — COVID-19; Anosmia | interventions — Smell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RT-PCR SARS-CoV-2 positive
  Interventions: Other: olfactory and gustatory tests
- RT-PCR SARS-CoV-2 negative
  Interventions: Other: olfactory and gustatory tests

INTERVENTIONS:
Other: olfactory and gustatory tests — Participants rate quality of sense of smell and taste.
  Olfaction test: Sniff 10ml test tube containing 1.5ml air freshner (Mifleur Citron, Coldis, Entraigues sur Sorgues, France) and rate perception of odor.
  Gustatory test: Taste a pinch and sugar and salt and rate perception of sweet or salty taste

SUMMARY:
Loss of sense of smell and taste has been anecdotally reported during the covid-19 epidemic. The study investigators wanted to describe the prevalence of olfactory and gustatory dysfunction and assess the factors associated with positive SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with COVID-19 related symptoms including: fever, persistent cough, fatigue, shortness of breath, diarrhoea, abdominal pain, chest pain, sore throat, loss of smell or taste
* Subjects in prolonged contact with COVID-19 infected patients.

Exclusion Criteria:

* Patients directly admitted to the intensive care unit were excluded
* Patients opposing use of their health data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults referred for a suspicion of COVID-19 infection and tested by RT-PCR assay for detection of SARS-CoV-2 in a nasopharyngeal sample at the COVID Screening Center or in the infectious and tropical diseases department of the University Hospital of Nîmes,
Sampling Method: Non-Probability Sample
Enrollment: 454 (Actual)
Dates: Start 2020-03-27 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
SARS-CoV-2 infection status | Day 0
  Positive/negative according to RT-PCR assay
Olfactory and gustatory loss | Day 0
  Custom-designed questionnaire (28 questions pertaining to symptoms, sense of smell and taste)

SECONDARY OUTCOMES:
Ability to detect odor | Day 0
  Ability to smell 1.5ml air freshner on a 0-100 VAS scale
Ability to detect odor | Six months
  Ability to smell 1.5ml air freshner on a 0-100 VAS scale
Ability to detect salty taste | Day 0
  Ability to taste a pinch of table salt on a 0-100 VAS scale
Ability to detect salty taste | Six months
  Ability to taste a pinch of table salt on a 0-100 VAS scale
Ability to detect sweet taste | Day 0
  Ability to taste a pinch of sugar on a 0-100 VAS scale
Ability to detect sweet taste | Six months
  Ability to taste a pinch of sugar on a 0-100 VAS scale
Olfactory and gustatory loss | Day 7
  Custom-designed questionnaire (28 questions pertaining to symptoms, sense of smell and taste)
Olfactory and gustatory loss | Day 14
  Custom-designed questionnaire (28 questions pertaining to symptoms, sense of smell and taste)
Olfactory and gustatory loss | Day 30
  Custom-designed questionnaire (28 questions pertaining to symptoms, sense of smell and taste)
Olfactory and gustatory loss | Day 60
  Custom-designed questionnaire (28 questions pertaining to symptoms, sense of smell and taste)
Severity of infection according to hospitalization rate | End of study (six months)
  % patients hospitalized
Olfactory and gustatory loss | Six months
  Custom-designed questionnaire (28 questions pertaining to symptoms, sense of smell and taste)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Lallemant, Principal Investigator — CHU Nimes
Locations (1):
- CHU de Nimes, Nîmes, France